CLINICAL TRIAL: NCT05687864
Title: Single-center, Multiple-strength, Single-dose Phase I Clinical Trial to Evaluate the Effect of Polyglycan Superparamagnetic Ferric Oxide Injection on Cardiovascular Magnetic Resonance Imaging in Patients With Chronic Kidney Disease
Brief Title: Study of Polyglycan Superparamagnetic Ferric Oxide Injection on Cardiovascular Magnetic Resonance Imaging
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DJTCSCYHT-I-04
Record Dates: First submitted 2023-01-05; First posted 2023-01-18 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2022-11

CONDITIONS: Magnetic Resonance Imaging; Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Polysaccharide superparamagnetic ferric oxide injection (Experimental): Participants will receive one single dose of 1mg/kg or 2mg/kg or 3mg/kg or 4mg/kg or 5mg/kg of Polysaccharide superparamagnetic ferric oxide injection on Day 1.
  Interventions: Diagnostic Test: Polysaccharide superparamagnetic ferric oxide injection

INTERVENTIONS:
Diagnostic Test: Polysaccharide superparamagnetic ferric oxide injection — The polysaccharide superparamagnetic ferric oxide injection is a clinical diagnostic reagent

SUMMARY:
Polysaccharide super paramagnetic ferric oxide injection is an iron supplement developed for patients with iron deficiency anemia. Due to its characteristics, it has the potential to be a contrast agent. The DJTCSCYHT-I-04 study is a single-center, multiple-strength and single-dose phase I clinical study on cardiovascular MRI in patients with chronic kidney disease, aiming to investigate the effects and safety of multi-strength, single-dose at different time points, and to provide reference for clinical diagnosis and MRI enhancement.

ELIGIBILITY:
Inclusion Criteria:

* The subjects voluntarily joined the study, signed the informed consent, and the compliance was good.;
* Age: ≥18 years old (at the time of signing the informed consent), gender is not limited;
* Patients diagnosed with Chronic Kidney Disease (CKD, 2012 KDIGO Guidelines);
* Eastern Cooperative Oncology Group (ECOG) score 0~1; Expected survival ≥3 months;
* Serum ferritin ≤ 1000μg/L and transferrin saturation ≤ 50%;
* The major organs function are good and meet the following criteria:

  1. blood routine examination:

     1. Hemoglobin ≥ 90g/L
     2. Neutrophil count (NEUT) ≥1.5×109/L;
     3. Platelet count (PLT) ≥ 75×109/L;
  2. Biochemical examination should meet the following standards:

     1. Total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal (ULN);
     2. Alanine transferase (ALT), aspartate transferase (AST) and gamma glutamyltransferase (gamma-GGT) ≤ 3ULN;
  3. Left ventricular ejection fraction (LVEF) ≥50%.
* Women of reproductive age should agree to use effective birth control during the study period and for 6 months after the study, and have a negative serum-pregnancy test within 7 days prior to study enrollment; Men should agree that effective birth control must be used during the study period and for six months after the end of the study period.

Exclusion Criteria:

* Had or currently have malignant tumors within 3 years. The following three conditions were eligible for inclusion:

  1. patients with other malignancies treated with a single operation achieved continuous 5-year disease-free survival (DFS);
  2. Cured cervical carcinoma in situ, non-melanoma skin cancer, and superficial bladder tumors [Ta (non-invasive tumor), Tis (carcinoma in situ), and T1 (tumor infiltrating basal membrane)];
  3. The disease was stable as assessed by the investigators, and the concomitant drugs did not affect medication during the trial and follow-up period.
* Subjects with any severe and/or uncontrolled medical conditions, including:

  1. Poorly controlled hypertension (systolic blood pressure ≥150mmHg or diastolic blood pressure ≥100 mmHg) or poorly controlled hypotension (systolic blood pressure <90mmHg or diastolic blood pressure <60 mmHg);
  2. Have ≥ grade 2 myocardial ischemia or myocardial infarction and/or severe or malignant arrhythmias [including QTc ≥450ms in men, QTc ≥470ms in women] and/or ≥ grade 2 congestive heart failure [New York Heart Association (NYHA)];
  3. Active infection (≥NCI, CTC AE 5.0, Grade 2);
  4. Viral hepatitis, syphilis, HIV and other infectious diseases;
  5. A history of immunodeficiency, including acquired or congenital immunodeficiency diseases, or a history of organ transplantation;
  6. People who have epilepsy and require treatment.
* Research and treatment related:

  1. Patients with iron deficiency anemia;
  2. Subjects who are allergic to intravenous iron preparations, the investigational drug or any of its components, or two or more types of drugs;
  3. Subjects who plan to undergo magnetic resonance imaging during the study period and during follow-up.
* Participants who have participated in other clinical trials of drugs or medical device within 28 days before the start of the study treatment;
* Those who have a history of psychotropic drug abuse and cannot abstain or have mental disorders;
* Pregnant or lactating women;
* Patients with non-magnetic compatible metal foreign bodies (false teeth, contraceptive rings, metal implants, metal clips, etc.) and claustrophobia; Patients with difficulty or inability to tolerate MRI scanning;
* Subjects with concomitant diseases that, in the investigator's judgment, seriously endanger subjects' safety or interfere with the completion of the study, or who are deemed unsuitable for enrollment for other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-06-17 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Signal-to-Noise Ratio (SNR) | Before administration, 5minutes, 24 hours, 48 hours after administration
  On the basis of vascular segments, the signal-to-noise ratio at different doses and time points was calculated by magnetic resonance imaging.
Contrast to noise ratio (CNR) | Before administration, 5minutes, 24 hours, 48 hours after administration
  On the basis of vascular segments, the Contrast to noise ratio at different doses and time points was calculated by magnetic resonance imaging.
Image quality score before administration | Before administration
  On the basis of vascular segments, the image quality of different doses at different time points was evaluated by magnetic resonance imaging. 4 points: the blood vessel edge is clear and sharp, without image artifacts, which can support the judgment of high confidence; 3 points: The overall portrayal effect of blood vessels was satisfactory, the anatomical structure of blood vessels was clear enough to meet the requirements of disease diagnosis, and there were mild image artifacts; 2 points: Blood vessels were visible, but only the local structure size or blood vessel patency could be judged, with moderate image artifacts;
  1 point: poor image quality, serious image artifacts, unable to distinguish blood vessels and other tissues, unable to evaluate.
Image quality score at 5 minutes | 5 minutes after administration
  On the basis of vascular segments, the image quality of different doses at different time points was evaluated by magnetic resonance imaging. 4 points: the blood vessel edge is clear and sharp, without image artifacts, which can support the judgment of high confidence; 3 points: The overall portrayal effect of blood vessels was satisfactory, the anatomical structure of blood vessels was clear enough to meet the requirements of disease diagnosis, and there were mild image artifacts; 2 points: Blood vessels were visible, but only the local structure size or blood vessel patency could be judged, with moderate image artifacts;
  1 point: poor image quality, serious image artifacts, unable to distinguish blood vessels and other tissues, unable to evaluate.
Image quality score at 24 hours | 24 hours after administration
  On the basis of vascular segments, the image quality of different doses at different time points was evaluated by magnetic resonance imaging. 4 points: the blood vessel edge is clear and sharp, without image artifacts, which can support the judgment of high confidence; 3 points: The overall portrayal effect of blood vessels was satisfactory, the anatomical structure of blood vessels was clear enough to meet the requirements of disease diagnosis, and there were mild image artifacts; 2 points: Blood vessels were visible, but only the local structure size or blood vessel patency could be judged, with moderate image artifacts;
  1 point: poor image quality, serious image artifacts, unable to distinguish blood vessels and other tissues, unable to evaluate.
Image quality score at 48 hours | 48 hours after administration
  On the basis of vascular segments, the image quality of different doses at different time points was evaluated by magnetic resonance imaging. 4 points: the blood vessel edge is clear and sharp, without image artifacts, which can support the judgment of high confidence; 3 points: The overall portrayal effect of blood vessels was satisfactory, the anatomical structure of blood vessels was clear enough to meet the requirements of disease diagnosis, and there were mild image artifacts; 2 points: Blood vessels were visible, but only the local structure size or blood vessel patency could be judged, with moderate image artifacts;
  1 point: poor image quality, serious image artifacts, unable to distinguish blood vessels and other tissues, unable to evaluate.

SECONDARY OUTCOMES:
T2* value of Liver | Before administration, and day 28, day 60, day 90 after administration
  T2* signals in the liver were quantitatively detected by magnetic resonance scanning
R2 value of Liver | Before administration, and day 28, day 60, day 90 after administration
  R2 signals in the liver were quantitatively detected by magnetic resonance scanning
Magnetic sensitivity of brain tissue | Before administration, and day 28, day 60, day 90 after administration
  Magnetic resonance scanning was used to quantitatively detect magnetic sensitivity of brain tissue
Incidence of adverse events | From the enrollment of the subjects to 90 days after administration
  The incidence of adverse events as assessed by Common Terminology Criteria for Adverse Events (CTCAE v5.0)
Incidence of severe adverse events | From the enrollment of the subjects to 90 days after administration
  The incidence of severe adverse events as assessed by Common Terminology Criteria for Adverse Events (CTCAE v5.0)

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Chaoyang Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No